CLINICAL TRIAL: NCT06483711
Title: Reducing Barriers to Lifestyle Modification for Pediatric Patients of Hispanic Ethnicity and Newly Diagnosed MASLD
Brief Title: Reducing Barriers to Lifestyle Modification for Newly Diagnosed MASLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rachel Herdes, CLINICAL ASSISTANT PROFESSOR, PEDIATRICS - GASTROENTEROLOGY, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-75991
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Lifestyle Kit Group (Experimental): Participants will receive a healthy lifestyle kit and be asked interview questions about its efficacy.
  Interventions: Other: Lifestyle Kit

INTERVENTIONS:
Other: Lifestyle Kit — The investigators will provide a kit to families that contains educational information, exercise equipment, and nutritional products.

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is the most common cause of liver disease in the world. It is estimated that 38% of American children with obesity have steatotic liver disease. Patients of Hispanic ethnicity are disproportionately at risk of developing MASLD. This study intends to provide insight to barriers of recommended care for pediatric patients with Hispanic ethnicity and a new diagnosis of MASLD. The investigators propose to augment existing structural barriers related to health literacy, food accessibility and dietary knowledge, and access to safe physical activity through a healthy lifestyle toolkit and individualized nutritional counseling.

DETAILED DESCRIPTION:
The Hispanic population represents the largest and fastest growing ethnic group in the United States. Patients of Hispanic ethnicity are disproportionately at risk of developing MASLD. An adult meta-analysis found a prevalence rate of 22.9% among individuals of Hispanic ethnicity. A pediatric retrospective study found that children who are Hispanic are 5 times more likely to have MASLD than their age/gender matched peers who identify as black. The etiology of why individuals of Hispanic ethnicity are at higher risk of developing MASLD, and subsequently associated co-morbidities such as insulin resistance, diabetes, and cardiovascular disease, is thought to be multifactorial. There is evidence to suggest that individuals of Hispanic ethnicity have a genetic predisposition for hepatic fat infiltration.11 Additionally, it has been postulated that social determinants of health, such as economic stability and health care access and quality contribute to an increased risk.

The American Association for the Study of Liver Diseases (AASLD) recommends lifestyle modification as the foundation of treatment for MASLD. Implementing dietary changes and increasing physical activity contribute to weight loss, which has been found to reduce hepatic steatosis. A 7-10% weight loss can improve histopathological features of MASLD, including fibrosis.Application of dietary modification, such as adherence to the Mediterranean dietary pattern, can decrease hepatic fat content, even in the absence of weight loss.Though lifestyle intervention has been found to be effective, barriers to implementation exist. In a study of adult patients of Hispanic ethnicity with a diagnosis of MASLD, access to nutritious food and a safe exercising environment limited the ability to follow through with recommended lifestyle changes.A survey study of pediatric patients with MASLD found that many lacked the opportunity for physical activity, though the majority expressed an interest in participation.16 Health literacy, or the ability to obtain and comprehend medical information, has also been found to be a barrier to effective care. In a qualitative interview study of adults with MASLD, health literacy was hindered by the availability of liver disease resources in the patient's preferred language. There is limited pediatric data regarding perceived barriers to implementing lifestyle changes. With this study, the investigators hope to minimize some of the social determinants of health that can impact Hispanic pediatric MASLD patients and help them participate in the recommended standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adolescent patients age 10-17 years of Hispanic ethnicity and newly diagnosed MASLD (as confirmed by ultrasound or biopsy + cardiometabolic risk factor) in the pediatric hepatology or GI clinic. Patients will also be restricted to patients who live in Alameda, Contra Costa, Solano, San Francisco, San Mateo, and Santa Clara counties due to the limitations of Fresh Approach locations. Families that include one family member who speaks English.

Exclusion Criteria:

* Age less than 10 and age greater than 17. Patient who do not live in Alameda, Contra Costa, Solano, San Francisco, San Mateo, and Santa Clara counties due to limitations of Fresh Approach locations. Families with no English Speakers or families whose primary language is not English or Spanish.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Social Determinants of Health Impacting Participants | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  Social Determinants of Health Screener will identify the presence of food, housing, and/or transportation insecurity.

SECONDARY OUTCOMES:
Mean Change from Baseline AST at 3 or 6 month follow-up appointment | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  AST lab value
Mean Change from Baseline ALT at 3 or 6 month follow-up appointment | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  ALT Lab value
Mean Change from Baseline GGT at 3 or 6 month follow-up appointment | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  GGT Lab value
Mean BMI Change from Baseline at 3 or 6 month follow-up appointment | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  BMI
Mean Weight Change from Baseline at 3 or 6 month follow-up appointment | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  weight
Socioeconomic status of Participants participating in the study | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  Socioeconomic status
Ethnic background of Participants participating in the study | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  ethnic background
Primary language of Participants participating in the study | Baseline and month 3 or 6 depending on when the participant's follow up appointment with the physician is scheduled.
  primary language

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Herdes, DO, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No
There currently are no plans to share IPD.